CLINICAL TRIAL: NCT01132404
Title: A Phase 1/2, Open Label Study in Men With Prostate Cancer to Assess the Safety. Pharmacokinetics and Testosterone-Lowering Efficacy of TAK-448, Administered as a 1-Month Depot, Including a Randomized Portion With a Group Administered Leuprorelin
Brief Title: Study in Men With Prostate Cancer to Assess the Safety, Pharmacokinetics and Testosterone-Lowering Efficacy of TAK-448
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Developing new formulation of study drug. New study to open next year under a new protocol.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C18002; 2009-017668-18 (EudraCT Number)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; metastin (46-54), acetyl-tyrosyl(46)-hydroxypropyl(47)-threonyl(49)-azaglycyl(51)-methylarginyl(53)-tryptophyl(54)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-448 Dose 1 (Experimental)
  Interventions: Drug: TAK-448
- TAK-448 Dose 2 (Experimental)
  Interventions: Drug: TAK-448
- Leuprorelin (Active Comparator)
  Interventions: Drug: Leuprorelin

INTERVENTIONS:
Drug: Leuprorelin — Phase 2 portion of study: patients randomized to this arm will receive a subcutaneous injection of depot Leuprorelin in the abdomen once per month for up to 6 months
  Arms: Leuprorelin
Drug: TAK-448 — Phase 1 portion of study:
  Patients will be administered a single dose of depot formulation TAK-448 via subcutaneous abdominal injection and a single dose of placebo at a contralateral injection site
  Phase 2 portion of the study:
  Patients randomized to this arm will be administered depot formulation TAK-448 (up to 2 dose levels) via subcutaneous injection in the abdomen once per month for up to 6 months
  Arms: TAK-448 Dose 1; TAK-448 Dose 2

SUMMARY:
The phase 1 portion of this study is an open-label, multicenter, dose-escalation study of 1-month depot TAK-448 in adult males with prostate cancer who are either on gonadotropin releasing hormone (GnRH) therapy or who might be eligible for GnRH therapy in the future. The phase 2 portion of this study is an open-label, multicenter, randomized study in men with prostate cancer that will confirm the testosterone- and prostate specific antigen (PSA)- lowering potential of up to 2 dose levels of 1-month depot TAK-448.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Male 40 to 72 years of age
* Histologically-confirmed adenocarcinoma of the prostate having completed primary local treatment at least 6 months prior to screening
* Meet all laboratory evaluation values at screening as specified in protocol
* For phase 1 of the study only: Concurrent gonadotropin releasing hormone (GnRH) therapy with generally indolent or stable disease OR a potential candidate of GnRH at some time in the future. Patients with metastatic disease must be asymptomatic with only bone scan positive evidence of metastases. Patients with recurrent local disease will be asymptomatic without bladder, bowel or obstructive symptoms
* For phase 2 portion of the study only: evidence of progressive prostate cancer, which in the opinion of the referring physician and/or study investigator warrants the initiation of GnRH analog therapy. Such patients may have either elevated or rising PSA at least 6 months following primary local therapy (ies) or have evidence of metastatic disease not previously treated with GnRH analog therapy.
* Provision of informed consent and for the phase 1 portion of the study only, willing to participate with no expectation of therapeutic benefit
* Generally fit medical condition, with no acute or chronic medical conditions other than prostate cancer, affecting 2-year life expectancy
* Ability to understand and comply with protocol requirements
* Agreement to, even if surgically sterilized but not surgically castrated, practice effective barrier contraception OR abstain from heterosexual intercourse
* Suitable venous access for blood sampling

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in either the phase 1 or phase 2 portion of the study:

* Advanced or symptomatic metastatic prostate cancer requiring immediate GnRH or additional hormone therapy or requiring chemotherapy
* History of surgical castration
* History of nonskin cancer, other than prostate cancer, requiring active treatment within 2 years of screening
* History of cardiac surgery, within the previous 6 months or any planned elective surgeries, other than skin surgery, during the ensuing 6 months
* Compromise of bone marrow function that would reduce tolerance to repeated blood draws
* History of osteoporosis, unless actively controlled with treatment, or history of vertebral or femoral fracture within the past year
* History of seizures or currently on anticonvulsant medications
* History of major psychiatric illness (diagnosed psychosis or psychiatric illness requiring hospitalization)
* History of drug or significant alcohol abuse
* Participation in clinical trials or receipt of experimental therapy within 2 months of screening
* Serious infection within 14 days before first dose of study drug
* Known history of human immunodeficiency (HIV) infection, hepatitis B, or hepatitis C infection
* History of significant cardiovascular condition

In addition, for the phase 2 portion of the study, patients must not have any of the following exclusion criteria:

* Participation in the phase 1 portion of the study
* Prior or current use of a GnRH analog or androgen receptor antagonist as first-line hormone therapy (other than as neoadjuvant/adjuvant use)
* History of use of GnRH analog or antagonist (as adjuvant or neoadjuvant therapy) within the 6 months prior to screening
* History of known or documented primary failure of GnRH analog therapy
* History of rising PSA or disease progression while on a GnRH analog or combined androgen blockade (CAB) therapy

Ages: 40 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
For Phase 1 portion of study: to assess the safety and pharmacokinetics (PK) of TAK-448 in patients receiving a single dose of 1-month depot TAK-448 | 3 months
  Vital signs; 12-lead ECG; Clinical laboratory test results; Injection site-related skin reactions; Adverse Events (AEs)and Serious Adverse Events (SAEs); Maximum observed plasma concentration; Area under the plasma TAK-448 disposition curve; The time of last quantifiable concentration
For Phase 2 portion of study: to assess the safety and PK of TAK-448 and effect of TAK-448 on serum testosterone concentrations in patients receiving repeated doses of 1-month depot TAK-448 | 8 months
  Vital signs; 12-lead ECG; Clinical laboratory test results; Injection site-related skin reactions; Adverse Events (AEs)and Serious Adverse Events (SAEs; Area under the plasma TAK-448 disposition curve; trough plasma concentration; Serum testosterone concentration; proportion of patients with serum concentration below castrate level

SECONDARY OUTCOMES:
For Phase 1 portion of study: to assess the effect of 1-month depot TAK-448 on serum testosterone and luteinizing hormone (LH) concentrations in patients not receiving concomitant gonadotropin releasing hormone (GnRH) analog therapy | 3 months
  Serum testosterone and LH concentrations; proportions of patients with serum testosterone concentrations below castrate-level
For Phase 2 portion of study: to assess the effect of 1-month depot TAK-448 on serum prostate specific antigen (PSA) concentration | 8 months
  Serum PSA concentration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Hôpital Edouard Herriot, 5, Place d'Arsonval, Pavillon V - Urologie et chirurgie de la transplantation, Lyon, France